CLINICAL TRIAL: NCT00466570
Title: Prospective Randomized Comparison of Zymar(Gatifloxacin) and Vigamox (Moxifloxacin) in Killing Conjunctival Bacterial Flora Following a One-hour
Brief Title: Prospective Randomized Comparison of Zymar(Gatifloxacin) and Vigamox (Moxifloxacin) in Killing Conjunctival Bacterial Flora Following a One-hour Application
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Ta, Principal Investigator, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 8924
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Conjunctical Flora
MeSH Terms: interventions — Gatifloxacin; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gatifloxacin, moxifloxacin

SUMMARY:
Topical ophthalmic antibiotics are common prescribed just prior to eye surgery to lower the risk of infection. Previous studies have suggested that antibiotics containing a preservative (Zymar) kill bacteria much quicker than those without a preservative (Vigamox). The purpose of this research is to compare how quickly to the two commonly prescribed antibiotics eliminate bacteria from the eye surface.

ELIGIBILITY:
Inclusion Criteria:

* Age- older than 50 years of age
* Diagnosis- Cataract or had cataract surgery

Exclusion Criteria:

* Systemic or topical antibiotic treatment within 30 days
* Use of systemic or topical steroids
* Active ocular infection
* Ocular surgery in the past 6 months
* Allergy to fluoroquinolones

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04

PRIMARY OUTCOMES:
Antibiotic killing of conjunctival bacterial flora 1 hour after application

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ta, MD, Principal Investigator — Stanford University

REFERENCES:
- [Background] Ta CN, He L, Nguyen E, De Kaspar HM. Prospective randomized study determining whether a 3-day application of ofloxacin results in the selection of fluoroquinolone-resistant coagulase-negative Staphylococcus. Eur J Ophthalmol. 2006 May-Jun;16(3):359-64. PMID 16761235
- [Background] Mino de Kaspar H, Koss MJ, He L, Blumenkranz MS, Ta CN. Antibiotic susceptibility of preoperative normal conjunctival bacteria. Am J Ophthalmol. 2005 Apr;139(4):730-3. doi: 10.1016/j.ajo.2004.10.007. PMID 15808182
- [Background] de Kaspar HM, Kreidl KO, Singh K, Ta CN. Comparison of preoperative conjunctival bacterial flora in patients undergoing glaucoma or cataract surgery. J Glaucoma. 2004 Dec;13(6):507-9. doi: 10.1097/01.ijg.0000137872.19942.cf. PMID 15534478
- [Background] Ta CN, Chang RT, Singh K, Egbert PR, Shriver EM, Blumenkranz MS, Mino de Kaspar H. Antibiotic resistance patterns of ocular bacterial flora: a prospective study of patients undergoing anterior segment surgery. Ophthalmology. 2003 Oct;110(10):1946-51. doi: 10.1016/s0161-6420(03)00735-8. PMID 14522770
- [Background] Ta CN, Egbert PR, Singh K, Shriver EM, Blumenkranz MS, Mino De Kaspar H. Prospective randomized comparison of 3-day versus 1-hour preoperative ofloxacin prophylaxis for cataract surgery. Ophthalmology. 2002 Nov;109(11):2036-40; discussion 2040-1. doi: 10.1016/s0161-6420(02)01236-8. PMID 12414411